CLINICAL TRIAL: NCT02967406
Title: Impact of Lifestyle Modification on Prevention of Dementia, Chronic Kidney Disease, Diabetes, Chronic Obstructive Pulmonary Disease, Cancers and Cardiovascular Disease in a Thai General Population: Cluster Randomized Controlled Trial
Brief Title: Impact of Lifestyle Modification on the Development of Dementia, Chronic Kidney Disease, Diabetes, Chronic Obstructive Pulmonary Disease, Cancers and Cardiovascular Disease in a Thai General Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanpasitthiprasong Hospital (Other Government)
Collaborators: Dementia Association of Thailand (Unknown); Diabetes Association of Thailand (Unknown); The Endocrine Society of Thailand (Other); Nephrology Society of Thailand (Unknown); Thai Dietetic Society (Unknown); Ubon Ratchathani Public Health Office, Thailand (Other Government)
Responsible Party: Principal Investigator, P Chamnan, Principal Investigator, Sanpasitthiprasong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMR-571; HSRI 59-069 (Other Grant/Funding Number: Health System Research Institute); TCTR20161116001 (Registry Identifier: Thai Clinical Trials Registry); 59-00-0228 (Other Grant/Funding Number: Thai Health Promotion Foundation)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Dementia; Diabetes Mellitus; Chronic Kidney Disease; Cardiovascular Diseases; Malignancy; Chronic Obstructive Pulmonary Disease
Keywords: Lifestyle modification; Primary prevention; Community-based intervention; Randomized control trial
MeSH Terms: conditions — Dementia; Diabetes Mellitus; Renal Insufficiency, Chronic; Cardiovascular Diseases; Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle modification (Experimental): 4 x 4 lifestyle modification intervention, addressing four health behaviors including physical activity, diet, smoking and alcohol drinking, at four different levels, i.e. individual, household, group/ knowledge management, and community levels
  Interventions: Behavioral: 4 x 4 lifestyle modification
- Control (No Intervention): No special intervention will be given. Prevention and treatment in normal practice is allowed

INTERVENTIONS:
Behavioral: 4 x 4 lifestyle modification — Participants in the intervention group will be given 4x4 lifestyle modification intervention, which will address four health behaviors (diet, physical activity, alcohol drinking and smoking) at four different levels: individual, household, knowledge management and community levels. A new computer program called 'iActive' adapted from the GPAQ with add-on functions to allow real-time assessment and presentation of the energy expenditure along with recommendations specific to each individual will be used. Dietary counseling will be given individually following assessment using a new dietary assessment program called Dietary Assessment Scanning Calculator. Home visit will be done every 3 months by responsible nurses and village health volunteers. Knowledge management will be done through meetings between participants and villages with support from trained nurses. Situation analysis and community action will be encouraged to address four health behaviors.
  Arms: Lifestyle modification

SUMMARY:
This is a community-based cluster randomized control trial aimed to investigate the impact of lifestyle modification (diet, physical activity, alcohol drinking and smoking) on the development of dementia, diabetes, chronic kidney disease, cancers, chronic obstructive pulmonary disease and cardiovascular disease in an intermediate risk population in mixed urban-rural areas of Ubon Ratchathani.

DETAILED DESCRIPTION:
This is a community-based cluster randomized control trial aimed to investigate the impact of lifestyle modification (diet, physical activity, alcohol drinking and smoking) on the development of dementia, diabetes, chronic kidney disease, cancers, chronic obstructive pulmonary disease and cardiovascular disease in an intermediate risk population in mixed urban-rural areas of Ubon Ratchathani.

Objectives:

1. examine the impact of lifestyle modification on the development of dementia, diabetes, chronic kidney disease, cancers, chronic obstructive pulmonary disease and cardiovascular disease in an intermediate risk population in Ubon Ratchathani
2. examine the economic impact of lifestyle modification on prevention of dementia, diabetes, chronic kidney disease, cancers, chronic obstructive pulmonary disease and cardiovascular disease in an intermediate risk population in Ubon Ratchathani

Study design: community-based cluster randomized control trial

Setting: 60 villages randomly selected from mixed urban-rural areas in 15 districts of Ubon Ratchathani province.

Study population: 3,600 apparently healthy men and women aged 45-75 years who have resided in the village selected for at least one year. 4,000 men and women will be approached and screened.

Screening and baseline assessment:

After community consent, potential participants will be informed about the details of the project. For those who are willing to participate, written informed consent will be given before carrying out all research procedures. Participants will be questioned about their demographic characteristics, medical and family history, health behaviours including diet, physical activity, alcohol drinking and smoking. Physical activity will be assess using the Global Physical Activity Questionnaire (GPAQ) and diet will be assessed using 24 hour food recall. Their cognitive function will be assessed using the Mini-Mental State Exam (MMSE), Thai version, and clock drawing test and depression test will also be performed. Physical examination includes weight, height, blood pressure, waist and hip circumference as well as physical fitness test.

Fasting blood samples will be collected for the following laboratory tests: Complete blood count, creatinine, estimated glomerular filtration rate (eGFR), fasting plasma glucose, glycated haemoglobin (HbA1c), total cholesterol, triglyceride, HDL and estimated LDL-cholesterol, serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), thyroid stimulating hormone (TSH), Ca++, PO4-, urine creatinine/albumin, urine sodium & potassium.

Interventions:

Participants in 30 villages in the intervention group will be given 4x4 lifestyle modification intervention, which will address four health behaviors (diet, physical activity, alcohol drinking and smoking) at four different levels: individual, household, knowledge management and community levels. A new computer program called 'iActive' will be used. The program was adapted from the GPAQ with add-on functions to allow real-time assessment and presentation of the energy expenditure along with recommendations specific to each individual. Dietary counseling will be given individually following assessment using a new dietary assessment program called Dietary Assessment Scanning Calculator (DISC). Home visit will be done every 3 months by responsible nurses and village health volunteers in order to assess and give simple counseling about health behaviors. Knowledge management will be undertaken through meetings and forums between participants and villages with support from trained nurses. Situation analysis and agreed community action will be encouraged to address community problems concerning four health behaviors. A combination of these intensive interventions will be given for 3 years.

Follow-up and outcome ascertainment:

Participants will be followed at 1, 2, 5 and 10 years after baseline assessment for the development of the outcomes of interest. In each follow-up, procedures identical to baseline assessment will be done.

Primary outcome: Incident dementia Incident dementia will be ascertained by a battery of screening test (MMSE, clock drawing and depression tests) and those with abnormal test results will be referred to neuro-medicine specialists at the regional hospital for further investigations and diagnosis.

Secondary outcomes:

1. Type 2 diabetes mellitus
2. chronic kidney disease
3. cancers
4. chronic obstructive pulmonary disease
5. cardiovascular disease
6. body mass index
7. waist circumference
8. blood pressure
9. Fasting plasma glucose
10. HbA1c
11. Lipids (total cholesterol, triglyceride, HDL and estimated LDL)

Tertiary outcomes:

1. MMSE scores or Cognitive decline
2. Alzheimer's disease
3. Physical activity levels
4. Dietary intake
5. prevalence of current smokers
6. prevalence of alcohol consumption

ELIGIBILITY:
Inclusion Criteria:

* Thai nationality
* Age 45-75 years
* Have resided in the Ubon Ratchathani's villages for at least 1 year
* Those giving written informed consent to participate in the research project

Exclusion Criteria:

* Known case of dementia, chronic kidney disease, diabetes, chronic obstructive pulmonary disease, cancers and cardiovascular disease
* Unable to communicate well in Thai
* Unable to move or get physical exercise
* Those at risk of having complications from performing physical exercise
* Those diagnosed with cancers of any system/ organ or those in the end of life period

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2016-03; Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dementia | 10 years
  Number of participants with dementia. Incident dementia will be diagnosed by medical specialists (Neuro-Med) following a battery of screening tests, including mini-mental state exam, depression and clock drawing tests.

SECONDARY OUTCOMES:
Type 2 diabetes mellitus | 3, 5 and 10 years
  Number of participants with type 2 diabetes mellitus. Diabetes mellitus is biochemically and clinically diagnosed.
Cardiovascular disease | 5 and 10 years
  Number of participants with cardiovascular disease. Clinical diagnosis of cardiovascular disease. Diagnostic information will be obtained from medical records review and service reimbursement data.
Cancers | 5 and 10 years
  Number of participants with cancers. Diagnostic information will be obtained from medical records review and service reimbursement data.
Chronic obstructive pulmonary disease | 5 and 10 years
  Number of participants with physician-diagnosed chronic obstructive pulmonary disease. Diagnostic information will be obtained from medical records review and service reimbursement data.
Mortality | 5 and 10 years
  All-cause mortality retrieved from death certificate database, which captures deaths nationwide, dates of death and related causes.
Blood sugar | 1, 2, 5 and 10 years
  Blood sugar assessed as fasting plasma glucose and glycated hemoglobin (HbA1c)
Blood lipids | 1, 2, 5 and 10 years
  Blood lipids include total, LDL- and HDL-cholesterol and triglyceride

OTHER OUTCOMES:
Physical activity levels | 1, 2, 5 and 10 years
  Physical activity levels assessed using the global physical activity questionnaire (GPAQ)
Diet | 1, 2, 5 and 10 years
  Diet assessed by 24 hour food recall
Prevalence of current smokers | 1, 2, 5 and 10 years
  Percentage of current smokers in the study samples
Prevalence of alcohol consumption | 1, 2, 5 and 10 years
  Percentage of those who report alcohol consumption
Cognitive function | 2, 5 and 10 years
  Cognitive function assessed by MMSE score

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Boongird, MD, Study Director — Dementia Association of Dementia; Parinya Chamnan, MD, PhD, Principal Investigator — Sanpasitthiprasong Hospital; Wannee Nitiyanant, MD, Principal Investigator — Siriraj Hospital; Wichai Aekplakorn, MD, PhD, Principal Investigator — Ramathibodi Hospital, Mahidol University; Chanida Pachotikarn, PhD, Principal Investigator — Thai Dietetic Society; Chaicharn Deerochanawong, MD, Principal Investigator — Rajvithi Hospital; Surasak Kantachuvesiri, MD, PhD, Principal Investigator — Ramathibodi Hospital, Mahidol University; Wallaya Jongjaroenprasert, MD, Principal Investigator — Ramathibodi Hospital, Mahidol University; Atiporn Ingsathit, MD, PhD, Principal Investigator — Ramathibodi Hospital, Mahidol University; Win Techakehakij, MD, PhD, Principal Investigator — Lampang Hospital; Phanida Krittayapoositpot, MD, Principal Investigator — Dementia Association of Thailand; Worawan Chailimpamontri, MD, Principal Investigator — Bhumibol Adulyadej Hospital; Ampika Mangklabruks, MD, Principal Investigator — Faculty of Medicine, Chiangmai University
Locations (1):
- Sanpasitthiprasong Hospital, Muaeng, Changwat Ubon Ratchathani, Thailand